CLINICAL TRIAL: NCT06138769
Title: Multicenter Phase 2 Trial of Lenvatinib in Patients With Unresectable or Metastatic Hepatocellular Carcinoma After Progression on First-line Atezolizumab Plus Bevacizumab
Brief Title: Lenvatinib After Progression on Atezolizumab-bevacizumab in Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Eisai Inc. (Industry); Chonnam National University Hospital (Other); Seoul National University (Other); Gangneung Asan Hospital (Other); Ulsan University Hospital (Other); Chosun University Hospital (Other); Dong-A University Hospital (Other); Bundang CHA Hospital (Other); Seoul National University Bundang Hospital (Other); Yonsei University (Other); Hanyang University Seoul Hospital (Other); Chungnam National University Hospital (Other); Saint Vincent's Hospital, Korea (Other); Gyeongsang National University Hospital (Other); Ewha Womans University (Other); Chungbuk National University Hospital (Other); Severance Hospital (Other); Gachon University Gil Medical Center (Other); The Catholic University of Korea (Other); Bucheon St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENVINEXT
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; lenvatinib; atezolizumab-bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib (Experimental): Lenvatinib 12 mg (body weight 60 kg or greater) or 8 mg (body weight < 60 kg) once orally every day
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 12 mg (body weight 60 kg or greater) or 8 mg (body weight < 60 kg) once orally every day

SUMMARY:
Although atezolizumab-bevacizumab has been positioned as the standard first-line therapy in unresectable heptocellular carcinoma, eventually most patients progressed on this regimen. Despite of multiple drugs are approved for the management of unresectable hepatocellular carcinoma, only a few trials have been conducted to investigate their efficacy in the second-line setting after the progression on atezolizumab-bevacizumab. Lenvatinib is approved first-line multikinase inhibitor in unresectable hepatocellular carcinoma, but has not yet been investigated as second-line therapy in prospective study. In this single arm phase 2 study, the efficacy and safety of lenvatinib will be investigated for patients who progressed on first-line atezolizumab-bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC according to AASLD guidelines
2. Disease that is not amenable to a curative treatment (e.g. surgery, transplant, radiofrequency ablation)
3. Prior treatment with atezolizumab plus bevacizumab as first-line treatment for unresectable HCC
4. Progression after atezolizumab plus bevacizumab, the duration of these treatments must be 2 consecutive treatment cycles or more.
5. At least 1 RECIST v1.1 measurable untreated lesion
6. Recovery to ≤ Grade 1 from toxicities related to any prior treatments, unless the adverse events are clinically non-significant and/or stable on supportive therapy
7. Life expectancy of 12 weeks or longer
8. Age ≥ 19 years old
9. ECOG performance status of 0, 1
10. Adequate hematological function

    1. Absolute neutrophil count (ANC) ≥ 1.0 x109/L
    2. Platelets ≥ 75 x 109/L
    3. Hemoglobin ≥ 10 g/dL
11. Adequate renal function

    1. serum creatinine ≤ 1.5 × upper limit of normal or calculated creatinine clearance ≥ 40 mL/min (using the Cockroft-Gault equation) AND
    2. urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.1 mg/mmol) or 24-hour urine protein < 1 g
12. Child-Pugh Score of 5 or 6
13. Total bilirubin ≤ 2 mg/dL (≤ 34.2 μmol/L)
14. Serum albumin > 2 g/dL (> 20 g/L)
15. Alanine aminotransferase (ALT) < 3.0 upper limit of normal (ULN)
16. Antiviral therapy per local standard of care if active hepatitis B (HBV) infection
17. Capable of understanding and complying with the protocol requirements and signed informed consent
18. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment
19. Females of child-bearing potential must be willing to use effective contraception during study and for 30 days after the last dose.

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. Prior lenvatinib treatment
3. Prior systemic treatment for HCC, except for atezolizumab plus bevacizumab (i.e. lenvatinib must be second-line systemic treatment)
4. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before randomization.
5. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders including i. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.

   ii. Uncontrolled blood pressure (Systolic BP>150 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.

   iii. Stroke (including TIA), myocardial infarction, or other ischemic event within 6 months iv. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.

   b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation/bleeding: i. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months
6. Major surgery within 2 months before randomization. Complete healing from major surgery must have occurred 1 month before randomization. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before registration. Subjects with clinically relevant co d. Cavitating pulmonary lesion(s) or endobronchial disease
7. Moderate or severe ascites (Radiologically detected but clinically insignificant ascites is allowed)
8. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 21 days of registration

   * If the QTcF is > 500 ms in first ECG, a total of 3 ECGs should be performed. If the average of these 3 consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard.
9. Subjects having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
10. Previously identified allergy or hypersensitivity to components of the study treatment formulations
11. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG [or hCG]).
12. Diagnosis of another malignancy within 2 years before randomization, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy
13. Electrolyte abnormalities that have not been corrected.
14. Subjects who have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy. Withhold lenvatinib for at least 1 week prior to elective surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing.
15. The participant has severe hypersensitivity (≥Grade 3) to lenvatinib and/or any of its excipients.
16. Other clinically significant disorders that are judged by investigators to be unsuitable for the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  Time interval between the start of lenvatinb to the disease progression or any cause of death.

SECONDARY OUTCOMES:
Overall survival | 1 year
  Time interval between the start of lenvatinib to the any cause of death
Overall response rate | 1 year
  Proportion of complete response or partial response according to the Response Evaluation Criteria for Solid Tumor version 1.1
Disease control rate | 1 year
  Proportion of complete response, partial response or stable disease according to the Response Evaluation Criteria for Solid Tumor version 1.1
Adverse events | 1 year
  Common Toxicity Criteria for Adverse Events version 5

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
It will be determined after the analysis of the primary data.

REFERENCES:
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Vogel A, Cervantes A, Chau I, Daniele B, Llovet JM, Meyer T, Nault JC, Neumann U, Ricke J, Sangro B, Schirmacher P, Verslype C, Zech CJ, Arnold D, Martinelli E; ESMO Guidelines Committee. Hepatocellular carcinoma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv238-iv255. doi: 10.1093/annonc/mdy308. No abstract available. PMID 30285213
- [Derived] Kim HD, Sym SJ, Chon HJ, Kim M, Kang JH, Ryoo BY, Lee CK, Hong J, Ryu H, Bae WK, Kim H, Kim H, Kim JW, Kim TY, Yoo C. Multicenter single-arm phase II trial of lenvatinib in patients with advanced hepatocellular carcinoma after progression on first-line atezolizumab plus bevacizumab. J Hepatol. 2026 Feb;84(2):308-315. doi: 10.1016/j.jhep.2025.08.020. Epub 2025 Sep 4. PMID 41038766